CLINICAL TRIAL: NCT03208192
Title: Comparison of Hydro-dissection Versus Ultrasonic Aspirator in Division of Liver Parenchyma in Laparoscopic Resection
Acronym: LLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Principal Investigator, Ivan Kazakov, Clinial Research, Moscow Clinical Scientific Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCNC 01/2017
Record Dates: First submitted 2017-06-26; First posted 2017-07-05 (Actual); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Liver Transection During Laparoscopic Liver Resection
Keywords: colorectal liver metastases; hepatocellular carcinoma; intrahepatic cholangiocellular carcinoma; tumor of liver; focal nodular hyperplasia liver; hemangioma liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: two groups will be compared. Group 1: liver resection using a bipolar dissector (Erbe), ultracision harmonic scalpel (Ethicon) and water-jet dissector (ERBEJET 2).
  Group 2: liver resection using a bipolar dissector (Erbe), ultracision harmonic scalpel (Ethicon), and ultrasonic aspirator (Misonix/SonaStar Ultrasonic Surgical Aspiration System)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ErbeJet (Experimental): liver resection using a bipolar dissector (Erbe), ultracision harmonic scalpel (Ethicon) and water-jet dissector (ERBEJET 2).
  Interventions: Procedure: liver transection during laparoscopic liver resection
- Misonix (Experimental): liver resection using a bipolar dissector (Erbe), ultracision harmonic scalpel (Ethicon), and ultrasonic aspirator (Misonix/SonaStar Ultrasonic Surgical Aspiration System)
  Interventions: Procedure: liver transection during laparoscopic liver resection

INTERVENTIONS:
Procedure: liver transection during laparoscopic liver resection — liver transection during laparoscopic liver resection

SUMMARY:
Background: until now, there is no agreement about the safest and feasible method for liver parenchyma transection during laparoscopic liver resection.

Study design: prospective, randomized, single-center The purpose of the study: comparison of short-term results of two methods of parenchyma liver transection during laparoscopic liver resection

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign lesions (hemangioma, focal nodular hyperplasia [FNH], hepatocellular adenoma, biliary cystadenoma, hydatid echinococcosis [only with total pericystectomy]) and malignant tumors (colorectal cancer metastases in the liver [CRLM], hepatocellular carcinoma [HCC], intrahepatic cholangiocellular carcinoma, gallbladder cancer T1b-3NxMo without invasion into bile ducts and adjacent organs), which involves laparoscopic segmental or major resection of the liver.
* Gender: both, male and female
* Minimum age 18 years
* Maximum age: 80 years
* ASA physical status I-IV
* BMI up to 40 kg/m2
* No simultaneous extrahepatic intra-abdominal procedures (bile duct resection, colon resection, partial duodenum resection)
* Total bilirubin up to 100mmol/l if jaundice presents in non-cirrhotic patients
* If cirrhosis is present, class A and B according to CTP score

Exclusion Criteria:

* • Difficulty index > 12 points (see below)

  * Tumor invasion of IVC or portal trunk (necessity of vascular reconstruction)
  * Repeated liver resection before laparoscopic resection (the single resection before is not a contraindication)
  * Simultaneous extra-hepatic intra-abdominal procedures (bile duct resection, colon resection etc.)
  * Age under 18 years
  * Age above 80 years
  * ASA physical status >IV
  * BMI > 40 kg/m2
  * Total bilirubin >100mmol/l if jaundice presents in non-cirrhotic patients
  * If cirrhosis is present, class C according to CTP score
  * Persons who are incapable of giving consent
  * Pregnant or breast-feeding women
  * Patients enlisted in other studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Efanov, MD, PhD, Study Chair — Moscow Clinical Scientific Center
Locations (1):
- Moscow Clinical scientific Center, Moscow, Entuziastov Shosse,86, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Partipants were recruited at Moscow Clinical Scientific Center. The first participant was enrolled on Feb 2017 and the last participant was enrolled in April 2020
Pre-assignment Details: Of 68 enrolled participants, met inlusion criteria and were randomized.
Period: Overall Study
Arm/Group | ErbeJet | Misonix
Started | 32 | 36
Completed | 32 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ErbeJet | Misonix | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 54 (15) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 12 | 15 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Median (Standard Deviation); unit: kg/m^2] | 28.4 (6.9) | 30 (5.2) | 29 (6.1)
Physical status classification system (ASA) [Count of Participants; unit: Participants] — ASA 1: A normal healthy patient. ASA 2: A patient with a mild systemic disease. ASA 3: A patient with a severe systemic disease that is not life-threatening. ASA 4: A patient with a severe systemic disease that is a constant threat to life. ASA 5: A moribund patient who is not expected to survive without the operation. The patient is not expected to survive beyond the next 24 hours without surgery. ASA 6: A brain-dead patient whose organs are being removed with the intention of transplanting them into another patient.
  Participants
    ASA 1 | 3 | 4 | 7
    ASA 2 | 15 | 20 | 35
    ASA 3 | 14 | 12 | 26
Malignant/benign lesions [Count of Participants; unit: Participants]
  Malignant | 18 | 24 | 42
  Bening | 14 | 12 | 26
Tumor size (mm) [Median (Full Range); unit: mm] | 71 [18 to 211] | 51 [16 to 165] | 61 [16 to 211]
Postero-superior segments [Count of Participants; unit: Participants] | 16 | 20 | 36
Difficulty index score (IWATE Criteria) Low\Intermediate\Advanced\Expert [Median (Full Range); unit: units on a scale] — IWATE criteria proposed at the International Consensus Conference on Laparoscopic Liver Resection as difficulty scoring system for laparoscopic liver resection. Difficulty index includes the type of liver resection (partial resection, segmentectomy, and sectionectomy), the size and topography of the tumor, its proximity to the large vessels of the liver, the presence and stage of liver cirrhosis (CTP) and has a scale ranging from 0 to 12. Difficalty level: low 0-4, intermediate 4-6, advanced 7-9, expert 10-12.
  units on a scale | 7 [2 to 12] | 7 [2 to 12] | 7 [2 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Blood Loss
Description: Absolute blood loss (ml) will be calculated as the amount of blood (collected only during the parenchyma resection) in suction the container after the subtraction of all irrigating fluids and weighing operative sponges.
Time Frame: 1 day
Measure: Mean (Full Range); unit: ml
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
ml | 195 [10 to 400] | 218 [10 to 1400]

2. Secondary Outcome: Аbsolute Measurement of Blood Loss in Relation to Resection Size (ml/cm^2)
Description: Аbsolute measurement of blood loss in relation to resection size (ml/cm^2).
Time Frame: 1 day
Measure: Mean (Full Range); unit: ml/cm^2
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
ml/cm^2 | 3.9 [0.9 to 10.6] | 5 [0.4 to 20]

3. Secondary Outcome: Duration of Liver Parenchyma Transaction
Description: Duration of liver parenchyma transaction (min)
Time Frame: 1 day
Measure: Median (Full Range); unit: min
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
min | 107 [19 to 305] | 100 [20 to 300]

4. Secondary Outcome: Necessity to Apply the Pringle Maneuver.
Description: the number of participants who needed to apply the Pringle maneuver
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
participants | 15 | 21

5. Secondary Outcome: The Total Duration of Pringle Maneuver.
Description: The total duration of Pringle maneuver (min)
Time Frame: 1 day
Measure: Median (Full Range); unit: min
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
min | 23 [3 to 59] | 18 [2 to 48]

6. Secondary Outcome: Hospital Stay (Day)
Description: Hospital stay (day)
Time Frame: up to 1 month
Measure: Mean (Full Range); unit: day
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
day | 8 [5 to 16] | 8 [4 to 19]

7. Other Pre Specified Outcome: Morbidity
Description: Morbidity according to Clavien-Dindo classification (it is advisable to activate complications class II-V). The Clavien-Dindo classification (CDC) is a standardized system for the registration of surgical complications. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The major characteristic of the CDC system is that the severity of a complication is graded based on the type of therapy required to treat the complication. The CDC system has been validated and accepted worldwide for use in many fields of surgery. The complications that change the treatment of grade II-V.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ErbeJet | Misonix
Number analyzed (Participants) | 32 | 36
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 30 days after the operation
Description: The definition of adverse event, used to collect adverse event information, no differs from the clinicaltrials.gov Definitions
Arm/Group | ErbeJet | Misonix
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/32 | 2/36
Other Adverse Events (participants affected / at risk) | 2/32 | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ErbeJet (N=32) | Misonix (N=36)
fluid accumulation (Hepatobiliary disorders) | 2 (2) | 2 (2) — postoperative fluid accumulation in the area of liver resection. Percutaneous puncture treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ErbeJet (N=32) | Misonix (N=36)
fluid collection (Surgical and medical procedures) | 2 (2) | 2 (2) — liquid accumulation along the line of liver resection that required percutaneous puncture

LIMITATIONS AND CAVEATS:
an addition to the exclusion criteria specified in the design of the study, the latter were expanded due to the following position. This made it difficult to recruit patients to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03208192/Prot_000.pdf
  • Informed Consent Form (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03208192/ICF_001.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT03208192/SAP_002.pdf